CLINICAL TRIAL: NCT06668610
Title: An Integrated Multifocal TDCS-EEG Protocol for Improving Cognitive and Affective Symptoms in Mild Cognitive Impairment and Early Stages of Dementia: a Crossover Double-blind Randomised Controlled Trial
Brief Title: A Multifocal TDCS-EEG Protocol for Improving Symptoms of Mild Cognitive Impairment and Early Dementia
Acronym: MuSt-MID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Luigi Trojano, Professor, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Vanvitelli_DeptPsy_30/2024
Record Dates: First submitted 2024-10-29; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Mild Cognitive Impairment (MCI); Dementia; Alzheimer Disease, Early Onset; Alzheimer Disease; Frontotemporal Degeneration (FTD); Neurocognitive Decline
Keywords: non invasive brain stimulation (NIBS); transcranial direct current stimulation (tDCS); electroencephalography (EEG); crossover; randomised controlled trial; mild cognitive impairment; early stage dementia; multifocal brain stimulation
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Alzheimer Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: The study will adopt a double-blinded crossover randomised controlled design. The whole intervention will consist of two treatment phases (sham vs real multifocal stimulation) and multiple assessment phases performed before and after each rehabilitation cycle (T1, T2, T3). Recruited participants will be randomly assigned to a "SHAM-REAL" stimulation group or a "REAL-SHAM" stimulation group by computer-generated random numbers. Throughout the entirety of the study, all participants will undergo conventional cognitive stimulation therapy, involving paper-and-pencil exercise and computerised activity on several cognitive domains including memory, attention, and executive functions (Bahar-Fuchs et al., 2019; Woods et al., 2012).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SHAM-REAL tDCS Group (Experimental): Participants randomly assigned to this group will receive a first cycle of SHAM multifocal tDCS (8 sessions, twice a week) and a second cycle of REAL multifocal tDCS (8 sessions, twice a week). During both cycles participant will receive cognitive stimulation treatment after brain simulation.
  Interventions: Device: StarStim 32, Neuroelectrics, Spain - Real multifocal tDCS; Device: StarStim 32, Neuroelectrics, Spain - Sham multifocal tDCS; Behavioral: Cognitive treatment
- REAL-SHAM tDCS Group (Experimental): Participants randomly assigned to this group will receive a first cycle of REAL multifocal tDCS (8 sessions, twice a week) and a second cycle of SHAM multifocal tDCS (8 sessions, twice a week). During the two cycles participant will receive cognitive stimulation treatment after brain simulation.
  Interventions: Device: StarStim 32, Neuroelectrics, Spain - Real multifocal tDCS; Device: StarStim 32, Neuroelectrics, Spain - Sham multifocal tDCS; Behavioral: Cognitive treatment

INTERVENTIONS:
Device: StarStim 32, Neuroelectrics, Spain - Real multifocal tDCS — Real multifocal tDCS will be delivered with an intensity of 2.0 mA over 8 electrodes positioned over the frontal and temporal areas in the left hemisphere according to the international 10/10 EEG system. The overall duration of stimulation will be set at 20 minutes.
  Other Names: transcranial Direct Current Stimulation
Device: StarStim 32, Neuroelectrics, Spain - Sham multifocal tDCS — Sham multifocal tDCS will be delivered with an intensity of 2.0 mA over 8 electrodes positioned over the frontal and temporal areas in the left hemisphere according to the international 10/10 EEG system. The overall duration of stimulation will be set at 30 seconds.
  Other Names: transcranial Direct Current Stimulation
Behavioral: Cognitive treatment — During the two cycles, all participants will undergo traditional cognitive stimulation therapy, involving paper-and-pencil exercise and computerised activity on several cognitive domains including memory, attention, and executive functions (duration 30-40 minutes) .

SUMMARY:
The goal of this clinical trial is to learn if an integrated protocol using multifocal non invasive brain stimulation and brain recording combined with cognitive training is effective in treating cognitive and affective symptomatology in patients with mild cognitive impairment and early stages of dementia. The main questions it aims to answer are:

* Does multifocal non-invasive brain stimulation reduce cognitive and affective symptoms in patients with mild cognitive impairment and early stages of dementia?
* Do some specific factors, such as education and cognitive reserve, affect the extent of the possible outcomes achievable from the intervention?
* Do electrophysiological measures contribute identifying responders and non-responders to the treatment? Researchers will compare real non-invasive brain stimulation to a placebo stimulation (reproducing the same feeling of stimulation without actually stimulating the brain) combined with cognitive rehabilitation on general cognition measures and depression symptoms.

Participants will

* Undergo two treatment cycles (real stimulation or placebo over frontal and temporal ares of the left hemisphere) combined with cognitive training twice a week for two months.
* Complete neuropsychological evaluations before the first rehabilitation cycle and at the end of each rehabilitation cycle.

Caregivers will provide information on functional daily living activities for their relatives.

DETAILED DESCRIPTION:
The global prevalence of dementia is expected to continue to rise. Recent estimates forecast that the number of people with dementia worldwide will increase to 152 million cases in 2050. This calls for the development of effective prevention and treatment strategies. Recently, the benefits of non-pharmacological interventions for the intervention in dementia and its preclinical conditions are being explored. Within this contex, transcranial direct current stimulation (tDCS), represents a safe and straightforward approach to modulate brain excitability with the potential to reduce symptomatology in individuals with dementia and Mild Cognitive Impairment (MCI).

The objective of this study is to evaluate a protocol for the treatment of the cognitive and affective symptoms in dementia and MCI with several specific novel features.

First, the protocol adopts multifocal stimulation of relevant brain structures involved in the genesis of the symptoms. While previous studies focused on specific areas in the frontal and temporal cortex in separate treatment conditions, the present study employes multifocal tDCS over such structures to strengthen distribution of direct current over the left fronto-temporal network, and to possibly boost the achievable outcomes.

Second, to address the issue of heterogeneity of stimulation effects, the study combines electrophysiological measures (EEG) with brain stimulation to monitor the effect of brain stimulation following specific polarities, also considering possible individual differences in response to stimulation. Such a protocol would allow identifying responders (and non responders) to stimulation, thus targeting individuals which may benefit (or not) from a given intervention.

Third, the study will further explore the variability in response to brain stimulation raised by previous studies, considering the relationship between some demographic and psychological factors with clinical and electrophysiological outcomes. Previous studies have shown a buffering effect of age and education on global cognitive response following brain stimulation, and a relevant association of cognitive functioning with cognitive reserve. The contribution of these variables will be explored in the study to provide a more complex interpretation of either positive or null effects associated with the intervention.

ELIGIBILITY:
Inclusion Criteria:

* age between 55 and 85 years;
* diagnosis of minor neurocognitive disorder, or major neurocognitive disorder with mild severity, according to Diagnostic and Statistical Manual of Mental Disorders (DSM-5; APA 2013) with a Clinical Dementia Rating Scale (CDR) of .05 or 1 (Morris, 1993);
* right handedness.

Exclusion Criteria:

* brain events with an acute aetiology (stroke, traumatic brain injury, neoplastic ablation);
* psychiatric disorders (schizophrenia, psychosis, bipolar disorder) and assumption of psychotropic drugs;
* diagnosis of moderate or severe major neurocognitive disorders (DSM-5; APA 2013) with CDR scores equal or above 2 (Morris, 1993);
* any condition with may also hypothetically interfere with electrophysiological recording and neurostimulation (metallic implants in the brain, cochlear implant, pacemakers, or suffering from epilepsy) (Antal et al., 2017; Bikson et al., 2016).

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MOCA; Santangelo et al., 2015). | The test will be used to monitor cognitive functions before the first cycle (T1, at week 0) and at the end of the first (T2; at week 4) and second cycle (T3; at week 8) of the intervention. Each cycle is 28 days.
  MOCA is a brief neuropsychological tool for screening global cognitive functioning specifically designed for MCI and early stages of dementia. The score ranges 0-30; the higher the score the higher the level of general cognitive functioning.
Frontal Assessment Battery (FAB; Appollonio et al., 2005). | The test will be used to monitor cognitive functions before the first cycle (T1, at week 0) and at the end of the first (T2; at week 4) and second cycle (T3; at week 8) of the intervention. Each cycle is 28 days.
  FAB is a screening neuropsychological battery for evaluation of executive functioning. Total score ranges 0-18; the higher the score, the higher the level of executive functioning.
Free and Cued Selective Reminding Test (FCSRT; Frasson et al., 2011). | The test will be used to monitor cognitive functions before the first cycle (T1, at week 0) and at the end of the first (T2; at week 4) and second cycle (T3; at week 8) of the intervention. Each cycle is 28 days.
  FCSRT is a neuropsychological tool designed to assess episodic memory domain. The test provides separate scores for free, cued and total immediate recall (scores 0-36), and scores for free, cued and total delayed recall (scores 0-12); the higher the scores, the higher the memory performance
Stroop Colour and Word Test (Caffarra et al., 2002). | The test will be used to monitor cognitive functions before the first cycle (T1, at week 0) and at the end of the first (T2; at week 4) and second cycle (T3; at week 8) of the intervention. Each cycle is 28 days.
  The Stroop Test is a neuropsychological test assessing cognitive interference and inhibition. The test provides two measures, i.e. overall number of errors and time to complete the test, with lower scores indicating better performance.
Geriatric Depression Scale (GDS; Galeoto et al., 2018). | The test will be used to monitor affective symptoms before the first cycle (T1, at week 0) and at the end of the first (T2; at week 4) and second cycle (T3; at week 8) of the intervention. Each cycle is 28 days.
  GDS is an evaluation tool to diagnose older adult's depression. This questionnaire is designed for the older person and defines his/her degree of satisfaction, quality of life, and feelings. The total score ranges 0-30 with higher scores indicating higher levels of depression.

SECONDARY OUTCOMES:
EEG Power Spectrum | EEG recordings will be performed before and after the first (at week 0), eight (at week 4), ninth (at week 5) and sixtheenth (at week 8) intervention sessions. The scale will be completed by caregivers. Each intervention cycle is 28 days.
  EEG data will be separated into two-second epochs after they are cleared of noise. Power spectrums of these data will be obtained in the delta, theta, alpha, beta and gamma frequency bands. Each epoch will be analyzed by Fast Fourier Transform (FFT, Fast Fourier Transform). Maximum peaks will be determined in the delta (0.5-3.5 Hz), theta (4-7 Hz), alpha (8-13 Hz), beta (15-28 Hz) and gamma (28-48 Hz) frequency bands. These values will be used in statistical analysis for each person and electrode.
Independence in Everyday Life - ADL | The scale will be used to monitor symptoms before the first cycle (T1, at week 0) and at the end of the first (T2; at week 4) and second cycle (T3; at week 8) of the intervention. The scale will be completed by caregivers. Each cycle is 28 days.
  Activities of Daily Living (ADL) Scale. The ADL refers to activities concerning care of one's own body, such as bathing, toileting, dressing and eating. The score ranges 0-6, with higher scores indicating higher levels of independence.
Independence in Everyday Life - IADL | The scale will be used to monitor independence before the first cycle (T1, at week 0) and at the end of the first (T2; at week 4) and second cycle (T3; at week 8) of the intervention. The scale will be completed by caregivers. Each cycle is 28 days.
  Instrumental Activities of Daily Living (IADL) Scale. The IADL refers to activities to support daily life within the home and community, such as financial management, housekeeping, shopping for groceries, making telephone calls, and taking medication. The score ranges 0-8, with higher scores indicating higher levels of independence.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology, University of Campania "Luigi Vanvitelli", Caserta, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Catalano L, Sagliano L, Visciglio A, Russo P, Miniello S, Trojano L, Panico F. An integrated multifocal tDCS-EEG protocol for reducing cognitive and affective symptoms in mild cognitive impairment and early stages of dementia: a crossover double-blind randomized controlled trial. Front Neurol. 2025 Jun 18;16:1605970. doi: 10.3389/fneur.2025.1605970. eCollection 2025. PMID 40606130